CLINICAL TRIAL: NCT00985127
Title: A Phase 2, Randomized, Double-Blind, Dose-Ranging, Two-Part, Multi-Center Study to Evaluate the Urate-Lowering Activity and Safety of Oral BCX4208 Administered in Subjects With Gout
Brief Title: Study to Evaluate the Urate-Lowering Activity and Safety of Oral BCX4208 Administered in Subjects With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX4208-201
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Gout
Keywords: Hyperuricemia; Gout
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — ulodesine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 40 mg (Experimental): 40 mg BCX4208
  Interventions: Drug: BCX4208
- 80 mg (Experimental): BCX4208
  Interventions: Drug: BCX4208
- 120 mg (Experimental): BCX4208
  Interventions: Drug: BCX4208
- sugar pill (Placebo Comparator)
  Interventions: Drug: placebo
- 160mg (Experimental): BCX4208
  Interventions: Drug: BCX4208
- 240mg (Experimental): BCX4208
  Interventions: Drug: BCX4208
- 320mg (Experimental): BCX4208
  Interventions: Drug: BCX4208

INTERVENTIONS:
Drug: placebo — administered daily for 21 days
  Arms: sugar pill
Drug: BCX4208 — Administered daily for 21 days.
  Arms: 120 mg; 160mg; 240mg; 320mg; 40 mg; 80 mg

SUMMARY:
The study will be conducted in two parts. The first is a parallel-group design, evaluating doses of 40 mg, 80 mg or 120 mg BCX-4208. The second part is planned as a dose-escalation study, evaluating higher doses including 160 mg, 240 mg and 320 mg BCX-4208. The study's primary endpoint is the change in uric acid in the blood compared to baseline measurement prior to treatment, assessed on Day 22.

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, double-blind study to evaluate the efficacy and safety of BCX4208 in approximately 120 subjects with gout. The study will be conducted in 2 parts. Part 1 is a parallel-group design, evaluating doses of BCX4208 previously found to be safe and well-tolerated in healthy subjects and subjects with psoriasis. Part 2 is a dose-escalation study, evaluating higher doses of BCX4208 supported by the nonclinical safety dossier. Part 2 will initiate after review of efficacy and safety data from Part 1, and determination that higher doses of BCX4208 may be necessary to achieve meaningful clinical activity.

In Part 1, approximately 60 subjects will be randomized in a 1:1:1:1 fashion to one of the following 4 treatment groups: 1) Placebo; 2) 40 mg BCX4208; 3) 80 mg BCX4208; or 4) 120 mg BCX4208.

In Part 1, the study will consist of 3 periods: the Screening Period, the Treatment Period, and the Follow-Up Period. The Screening period will begin on Day -30 for subjects receiving urate-lowering therapy; these subjects will discontinue the urate-lowering therapy on Day -30 to allow an appropriate washout period before entering the Treatment Period. For subjects not receiving urate-lowering therapy, the Screening Period may begin on any day from Day -30 to Day -1 (Day -1 being the day immediately prior to dosing), as long as all inclusion and exclusion criteria are satisfied.

Some Screening procedures such as a recording of medical history and some clinical laboratory tests (those that are performed at Screening only) may be performed at any time during the Screening Period (Day -30 to Day -1). Other Screening procedures must be performed within the 6 days prior to the first dose of study drug (i.e., from Day -6 to Day -1); these include: physical examination, height, weight, clinical chemistry (including baseline and qualifying sUA), hematology, and urinalysis evaluations, CD4+, CD8+, CD20+, and CD56+ lymphocyte counts, a serum pregnancy test, 12-lead electrocardiogram (ECG), and vital signs assessments. These assessments will constitute the Baseline assessments for the purpose of comparisons with these same assessments post-dose.

A recording of concomitant medications and adverse events (AEs) will take place from the time of the signing of the Informed Consent Form (ICF) and throughout the duration of the study.

The Treatment Period begins on Day 1. Subjects are to arrive at the study clinic on Day 1 after an overnight fast. After a final review of eligibility criteria, pre-dose vital signs assessments, and pre-dose BCX4208 pharmacokinetic (PK) blood draw have been performed, subjects will be randomized and administered the first dose of study drug. Subjects will remain in the study clinic for Hour 2, Hour 4, and Hour 8 assessments and will return to the study clinic for efficacy and safety evaluations on Days 2, 8, 15, and 22.

Subjects will take study drug daily from Day 1 to Day 21, so that the Day 22 evaluation will occur approximately 24 hours after the last dose of study drug.

After the Day 22 evaluation, subjects will enter the Follow-Up Period and will return to the study clinic on Days 29, 36, 43, and 50 for safety evaluations. Subjects who on Day 50 have unresolved treatment-emergent AEs will be followed beyond Day 50 until either resolution of the AE or until Day 80, whichever occurs sooner. Subjects who on Day 50 have absolute CD4+, CD8+, CD20+, and/or CD56+ lymphocyte counts that are both below the lower limit of normal and < 50% of Baseline will be followed monthly until the sooner of: 1) return of the absolute CD4+, CD8+, CD20+, and/or CD56+ lymphocyte counts to the lower limit of normal range, or 2) 6 months after the Day 50 or Early Termination Visit. All other subjects will conclude their study participation at the Day 50 or Early Termination Visit.

Efficacy will be assessed during the study by means of sUA concentrations. Safety will be assessed during the study by means of physical examination, weight, clinical chemistry, hematology, and urinalysis parameters, absolute CD4+, CD8+, CD20+, and CD56+ lymphocyte counts, 12-lead ECG, vital signs assessments, and AE assessments.

Efficacy, safety, and tolerability data from Part 1 of the study will be reviewed prior to initiation of Part 2.

Part 2 will consist of up to 3 cohorts: 1) 160 mg BCX4208 or placebo; 2) 240 mg BCX4208 or placebo; and 3) 320 mg BCX4208 or placebo. Unlike Part 1, Part 2 is a dose-escalation design whereby each of the cohorts will be enrolled sequentially, following review of the efficacy, safety, and tolerability data of the previous cohort. Enrollment into each cohort during Part 2 will be in a 3:1 ratio of BCX4208 to placebo such that 15 subjects will be randomized into each of the BCX4208 groups (total of 45 subjects) and 15 subjects will be randomized to placebo.

All study procedures for Part 2 of the study, from the Screening through the Follow-Up Period, will be conducted as described for Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 to <70 years
2. Have read and signed the ICF after the nature of the study has been fully explained
3. Screening sUA ≥8.0 mg/dL
4. Diagnosis of gout according to the preliminary criteria of the American Rheumatism Association (1977)
5. Female participants must meet at least one of the following specifications:

   * Be surgically sterile
   * Be post-menopausal as defined by:
   * females ≥55 years of age whose last menstrual period >1 year
   * females between ≥45 and <55 years of age whose last menstrual period > 1 year and FSH >40 mIU/mL and estradiol <40 pg/mL
   * Use oral contraceptives or some other form of hormonal birth control including hormonal vaginal rings or transdermal patches for 3 months prior to study drug dosing through 4 weeks after study drug administration
   * Use an intrauterine device as birth control for 8 weeks prior to study drug dosing through 4 weeks after study drug administration
   * Use (or ensure male partner[s]'s compliance with) a barrier contraception method (condom or diaphragm with a spermicide) for 4 weeks prior to study drug dosing through 4 weeks after study drug administration
6. Male participants must be considered not of child-bearing potential defined as >1 year post-vasectomy or use a condom for 4 weeks prior to study drug dosing through 4 weeks after study drug administration. In addition, they must ensure their sexual partner complies with the female contraception requirements specified above.
7. Be willing to avoid procreation for 3 months after study drug administration.
8. Be willing and able to provide authorization for the use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability policy.

Exclusion Criteria:

1. Unstable angina
2. History of cardiac arrhythmia
3. History of congenital long QT
4. Presence of cardiac signs or symptoms compatible with New York Heart Association Class III or Class IV functional status for congestive heart failure or angina
5. Uncontrolled hypertension (above 150/95 mm Hg)
6. History of moderate or severe renal impairment and/or previous clinical laboratory data indicating an estimated calculated creatinine clearance < 60 mL/min during the previous 12 months
7. ALT/AST values >2.0 x ULN
8. CD4+ cell counts by flow cytometry <500 cells/mm3 or >1600 cells/mm3
9. Hemoglobin <12 g/dL or >17 g/dL (males) or < 11 g/dL or >16 g/dL (females)
10. Hematocrit <37% or >51% (males) or <33 % or >47% (females)
11. WBC <3.7 x 109/L or >11 X 109/L
12. Immunocompromised due to illness or organ transplant
13. Current use of systemic immunosuppressive medications or treatments
14. Gout flare during the Screening Period that is resolved for less than 3 weeks prior to first treatment with study drug (exclusive of chronic synovitis/ arthritis)
15. Recipient of any live, attenuated vaccine within 6 weeks of Screening
16. History of clinically significant and relevant drug and/or food allergies
17. History of chronic or recurrent infections
18. History of any type of cancer (hematologic or solid tumor), that has required chemotherapy or radiation therapy in the previous 12 months, excluding non-melanomatous localized skin cancer
19. Use of uric acid-lowering drugs within 30 days prior to the first dose of study drug or other prohibited medications within the timeframes specified in the protocol
20. ACTH administration within 30 days of first treatment with study drug
21. Intra-articular corticosteroid administration within 30 days of first treatment with study drug
22. Systemic or oral glucocorticosteroid use within 4 weeks of first treatment with study drug or for a period of ≥ 6 months out of the last 12 months prior to the first treatment with study drug
23. History of alcohol or drug abuse within the year prior to the signing of the ICF, or current evidence of substance dependence or abuse (alcohol intake > 3 drinks per day)
24. Female subjects who are pregnant, planning a pregnancy or breastfeeding
25. Positive pregnancy test
26. Positive serology for hepatitis B or C surface antigen or human immunodeficiency virus (HIV) type 1
27. Have been the recipient of any investigational drug within the last 30 days prior to the first treatment with study drug
28. Other medical conditions which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject or impact the validity of the study results

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of different doses of orally administered BCX4208 on serum uric acid (sUA)levels in subjects with gout. | Day 22

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Radiant Research, Inc., Scottsdale, Arizona
  - Catalina Pointe Clinical Research, Tucson, Arizona
  - Irvine Center for Clinical Research, Irvine, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Avail Clinical Research, DeLand, Florida
  - Anchor Research Center, Naples, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Selah Medical Center, Boise, Idaho
  - Kentucky Medical Research Center, Lexington, Kentucky
  - Arthritis & Osteoporosis Center of Maryland, Frederick, Maryland
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Medex Healthcare Research, St Louis, Missouri
  - Bozeman Urgent Care Center, Bozeman, Montana
  - Heartland Clinical Research, Omaha, Nebraska
  - Arthritis Center of Reno, Reno, Nevada
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - STAT Research, Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Carolinas Center for Rheumatology & Arthritis, Rock Hill, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Renaissance Clinical Research, Dallas, Texas
  - Northwest Clinical Research Center, Bellevue, Washington